CLINICAL TRIAL: NCT06313515
Title: Transcutaneous Spinal Cord Stimulation Combined With Arm Crank Exercise for Cardiovascular Recovery in Cervical and Upper Thoracic SCI
Brief Title: Transcutaneous Spinal Cord Stimulation Combined With Arm Bike for Cardiovascular Recovery in SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Soshi Samejima, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00019529
Record Dates: First submitted 2024-03-03; First posted 2024-03-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries
Keywords: Transcutaneous Spinal Cord Stimulation; Arm-Bike Exercise; Cardiovascular Function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, sham-controlled trial with two arms (tSCS paired with arm-crank exercise compared to sham stimulation with exercise). Participants will be randomized into either the intervention or sham stimulation arm. Those in the sham arm only will initially receive sham stimulation, but then cross over to receive the active treatment arm, such that by the end all participants will have been exposed to the tSCS. tSCS participants will not receive sham stimulation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tSCS paired with arm-crank exercise (Experimental): Device: Transcutaneous Spinal Stimulation
  Non-invasive electrical stimulation of the spinal cord over the skin.
  Other: Arm-crank exercise
  Exercise using an arm-bike to target cardiovascular functioning.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation; Behavioral: Arm-crank bike exercise
- Sham stimulation paired with arm-crank exercise (Sham Comparator): Device: Sham Stimulation
  Non-invasive electrical stimulation of a lower extremity muscle group over the skin.
  Other: Arm-crank exercise
  Exercise using an arm-bike to target cardiovascular functioning.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation; Behavioral: Arm-crank bike exercise; Other: Sham Stimulation

INTERVENTIONS:
Device: Transcutaneous Spinal Cord Stimulation — Non-invasive electrical stimulation of the spinal cord over the skin
  Other Names: tSCS
Behavioral: Arm-crank bike exercise — Exercise using an arm-bike to target cardiovascular functioning.
  Other Names: arm-crank exercise
Other: Sham Stimulation — Non-invasive electrical stimulation of a lower extremity muscle group over the skin.
  Arms: Sham stimulation paired with arm-crank exercise

SUMMARY:
Spinal cord injury (SCI) can make it hard for the body to self-regulate some of its automatic functions like blood pressure, breathing, and heart rate. This can also make it hard for those living with SCI to exercise or complete their usual daily activities. The goal of this randomized trial is to test combinatory therapy of moderate arm-crank exercise paired with non-invasive transcutaneous spinal cord stimulation (tSCS) for cardiovascular recovery in adults aged 21-65 following chronic motor-complete spinal cord injury (SCI) at or above the thoracic sixth spinal segment (≥T6).

The main questions the study aims to answer are:

* Conduct tSCS mapping to determine the most effective location and stimulation intensity for BP control in individuals with motor-complete SCI ≥ T6.
* Evaluate the effects 8 weeks of targeted tSCS paired with arm-crank exercise compared to sham stimulation with exercise on improving cardiovascular function in individuals with motor-complete SCI ≥T6.
* Evaluate the dosage-response of 8 weeks vs. 16 weeks of targeted tSCS paired with arm-crank exercise on cardiovascular function in individuals with motor-complete SCI ≥T6.
* Explore the mechanisms involved in cardiovascular recovery with long-term tSCS paired with arm-crank exercise.

Participants will:

* Receive either transcutaneous spinal cord stimulation or "sham" spinal cord stimulation while exercising on an arm-crank bicycle in the first 8 weeks.
* Come in for approximately 60 visits over a 6-month period. This includes 2, 8-week periods where the investigators will ask participants to come in 3x per week for spinal cord stimulation and exercise.
* During assessment visits the researchers will perform a variety of exams including a neurologic, cardiovascular, pulmonary, physical, and autonomic exam, and will ask questions about quality of life and functioning.

Researchers will compare those who receive tSCS and do moderate arm-crank exercise to those who receive a sham stimulation and do moderate arm-crank exercise to see if tSCS is effective at improving cardiovascular and autonomic functioning in those with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Are between 21-65 years of age.
* Chronic SCI (non-progressive, with complete motor paralysis) at or above the T6 spinal cord segment.
* Greater than one year post injury or diagnosis, at least 6 months from any spinal surgery.
* American Spinal Injury Association Impairment Scale (AIS) A, B for SCI.
* Have stable medical condition without cardiopulmonary disease that would contraindicate participation in intensive training or testing activities.
* Cleared for strenuous exercise with arm bike by a primary physician of the subject (the clearance for intensive training with arm bike is obtained verbally or through a written form by a primary physician.)
* Willing and able to comply with all clinic visits and study-related procedures.
* Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
* Have no painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing.
* Are with stable management of spinal cord related clinical issues (i.e., spasticity management).
* Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

  -----Women of childbearing potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence.
* Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment.
* Are volunteering to be involved in this study.
* Has adequate social support to be able to participate in training and assessment sessions, up to 3 sessions per week, for the duration of up to 5 months within the study period.
* Must provide informed consent.

Exclusion Criteria:

* Have autoimmune etiology of spinal cord dysfunction/injury
* Have history of additional neurologic disease, such as stroke, MS, traumatic brain injury, etc.
* Have peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.)
* Have rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Are ventilator dependent.
* Have clinically significant, unmanaged, depression, ongoing alcohol and/or drug abuse.
* Use any medication or treatment that in the opinion of the investigators indicates that it is not in the best interest of the participant to participate in this study.
* Have Intrathecal baclofen pump.
* Have cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones.
* Have severe acute medical issue that in the investigators' judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to acute urinary tract infections, active heterotopic ossification, newly changed antidepressant medications [tricyclics], debilitating muscle pain, pressure sores, or unstable diabetes.
* Have pacemakers, stimulators, medication pumps in the trunk, deep brain stimulators, metallic devices in the head such as aneurysm clips/coils and stents, vagus nerve stimulators.
* Take more than 40 mg of Baclofen per day
* Have severe anemia (Hgb<8 g/dl or Hgb,80 g/L) or hypovolemia as measured by hematocrit via blood test in the last six months.
* Are a member of the investigational team or his/her immediate family.
* Have undergone electrode implantation surgery.
* Have signs of lower motor neuron impairment (i.e., concomitant conus medullaris/cauda equina injury).
* Have history of severe allergy (i.e. allergic reaction that could not be treated with antihistaminic medication)
* Have malabsorption syndrome, primary hyperthyroidism, and/or hypogonadism.
* Have a history of seizures.
* Have chronic headaches or migraines.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic Blood Pressure (BP) from baseline. | Baseline
  Continuous beat-by-beat BP will be measured using a finger photoplethysmography.
Change in systolic Blood Pressure during a sit-up test or head-up tilt test. | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Continuous beat-by-beat BP will be measured during a orthostatic challenge.
Heart rate variability recorded by electrocardiogram (ECG). | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Parameters using RR intervals (R-wave peak to R-wave peak in electrocardiogram) processed to assess the activity of autonomic nervous system.

SECONDARY OUTCOMES:
Peak oxygen uptake (VO2peak) | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Measured during incremental cardiopulmonary exercise test (CPET) on the arm-crank.
Autonomic dysfunction following Spinal Cord Injury (ADFSCI) measure | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  The Autonomic Dysfunction following SCI (ADFSCI) measure will be used to assess severity and frequency of autonomic dysreflexia. Greater scores equal greater frequency of autonomic dysfunction, ranging from 0 (never) to 4 (very often) for each item.
International Standards for Neurological Classification of Spinal Cord Injury | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  level and severity of damage to motor and sensory pathways will be determined by trained clinicians. Pin prick and light touch will be done by researchers on participant's left and right side. Check marks are given for each prick or touch that is felt by the participant, then tallied. Scores range from 0-56 for both the Left and Right side of the body, and 0-112 for the total score. High scores represent greater sensory functioning.
International Standards to document remaining Autonomic Function after Spinal Cord Injury (ISAFSCI) | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Scores for questions on the ISAFSCI range from 0 to 2, with 0 representing complete loss of control and 2 representing normal functioning. Lower scores equal worse health functioning.
Blood Pressure variability | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  BP Variability will be assessed using results from continuous beat-by-beat BP measurements obtained throughout the study using Finapres NOVA and a 24 hour BP monitoring assessment.
Change from baseline- Graded Redefined Assessment of Strength, Sensation, and Prehension version 2 | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Measurement of upper limb strength, sensation, qualitative prehension, and quantitative prehension (range 0-188, higher score mean better outcome)
Change from baseline- Capabilities of Upper Extremity Test | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Measures unilateral and bilateral hand and arm function (range 0-128, higher score mean better outcome)
International Spinal Cord Injury Pain Basic Dataset version 2.0 | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Standardized questionnaire for the collection and reporting of pain in the SCI population. Scores range from 0 to 10, with higher scores indicating greater pain interference and worse functioning.
International Spinal Cord Injury Lower Urinary Tract Function Dataset | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  The International SCI Lower Urinary Tract Function Dataset is a data collection form for the collection and reporting of lower urinary tract function in the SCI population. Participants are asked to mark either main or supplementary for type of bladder emptying, and then answer yes or no questions regarding type of appliances used to collect urinary incontinence, drugs with possible influence on urinary tract within the past 4 weeks, and any surgical procedures on the urinary tract. This data collection form does not use numbers and instead collects qualitative data only; there is no score range.
International Spinal Cord Injury Bowel Function Dataset | Repeated measurements before and after each 8 week-intervention block, an average of 6 months
  Standardized data collection form for the collection and reporting of bowel function in the SCI population. The International SCI Bowel Function Dataset is a data collection instrument that asks participants qualitative questions which are assigned a score. Select items are then totaled to compute the Neurogenic Bowel Dysfunction (NBD) score. Scores range from 0 to 14 or more, with higher scores indicating greater neurogenic bowel dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Soshi Samejima, DPT, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States